CLINICAL TRIAL: NCT02606682
Title: A Phase 1, Randomized, Double-Blind, Single Ascending Dose Trial of the Safety, Tolerability and Pharmacokinetics of NPT200-11 in Healthy Subjects
Brief Title: Phase 1 Study of NPT200-11 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuropore Therapies Inc. (Industry)
Collaborators: UCB S.A. - Pharma Sector (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPT200-11-001
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; Safety; Tolerability; Pharmacokinetics; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — NPT200-11; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- NPT200-11 - Cohort 1, Dose 1 (Experimental): Single ascending dose of orally administered capsule(s) NPT200-11: 15 mg OR Single dose of orally administered placebo capsule(s) to match dose
  Interventions: Drug: NPT200-11; Drug: Placebo
- NPT200-11 - Cohort 2, Dose 2 (Experimental): Single ascending dose of orally administered capsule(s) NPT200-11: 30 mg OR Single dose of orally administered placebo capsule(s) to match dose
  Interventions: Drug: NPT200-11; Drug: Placebo
- NPT200-11 - Cohort 3, Dose 3 (Experimental): Single ascending dose of orally administered capsule(s) NPT200-11: 60 mg OR Single dose of orally administered placebo capsule(s) to match dose
  Interventions: Drug: NPT200-11; Drug: Placebo
- NPT200-11 - Cohort 4, Dose 4 (Experimental): Single ascending dose of orally administered capsule(s) NPT200-11: 120 mg OR Single dose of orally administered placebo capsule(s) to match dose
  Interventions: Drug: NPT200-11; Drug: Placebo
- NPT200-11 - Cohort 5 ,Dose 5 (Experimental): Single ascending dose of orally administered capsule(s) NPT200-11: 240 mg OR Single dose of orally administered placebo capsule(s) to match dose
  Interventions: Drug: NPT200-11; Drug: Placebo
- NPT200-11 -Cohort 6, Dose 6 (Experimental): Single ascending dose of orally administered capsule(s) NPT200-11: 360 mg OR Single dose of orally administered placebo capsule(s) to match dose
  Interventions: Drug: NPT200-11; Drug: Placebo
- NPT200-11 - Cohort 7, Dose 7 (Experimental): Single ascending dose of orally administered capsule(s) NPT200-11: 480 mg OR Single dose of orally administered placebo capsule(s) to match dose
  Interventions: Drug: NPT200-11; Drug: Placebo

INTERVENTIONS:
Drug: NPT200-11 — Single doses of NPT200-11capsules, orally administered
Drug: Placebo — Single doses of microcrystalline cellulose capsules, orally administered
  Other Names: Microcrystalline cellulose capsules

SUMMARY:
The purpose of this study is to determine the safety, tolerability and blood levels of orally administered NPT200-11 in healthy subjects. In addition, the maximally tolerated dose will be determined.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following inclusion criteria will be eligible to participate in this study:

1. informed of, and willing and able to comply with, all of the protocol requirements and the investigational nature of the study, and have signed an informed consent form in accordance with institutional and regulatory guidelines;
2. male or female adults between 18 and 55 years of age, inclusive;
3. female subjects must be post-menopausal for at least 2 years or surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation);
4. male subjects must be willing to use an adequate barrier method of contraception for the duration of the study and for 90 days after dosing and no sperm donations for the duration of the study and for 90 days after dosing. Male subjects who are surgically sterile need not employ a method of contraception;
5. non-smokers for at least six months;
6. BMI = 18 - 30 kg/m2, inclusive;
7. in good health, in the judgment of the Principal Investigator, as determined by:

   * medical history indicative of no serious or severe chronic conditions requiring frequent medical intervention or continual pharmacologic management, and no medical or social conditions that would potentially interfere with the subject's ability to comply with the study visit schedule or the study assessments;
   * no clinically significant abnormalities in body temperature, heart rate, respiratory rate, blood pressure;
   * no clinically significant abnormalities in the 12-lead electrocardiogram (ECG);
   * no clinically significant abnormalities in clinical chemistry (ALT, AST, total bilirubin must be at or below the upper limit of normal and eGFR must be above 90 mL/min), hematology (hemoglobin ≥ 12.0 g/dL), coagulation and urinalysis; lab tests may be repeated, if necessary (details are provided in the attached flow chart of study assessments).
8. negative results on the following screening laboratory tests: urine drug screen, urine alcohol screen, serum pregnancy test, hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will NOT be eligible to participate in this study:

* females of child bearing potential;
* history of a significant medical condition that may interfere with absorption, distribution or elimination of NPT200-11, or with the clinical and laboratory safety assessments in this study;
* history of drug hypersensitivity and disorders affecting respiratory function (e.g., COPD, asthma) and cardiac disorders predisposing to cardiac adverse events;
* history of or current alcohol abuse and/or other drug addiction < 2 years prior to screening, or a positive urine drug or alcohol screen (e.g., amphetamines, barbiturates, benzodiazepines, opiates, cannabinoids, alcohol and cocaine);
* positive for HBVsAg, HCV Ab, HIV Ab;
* 12 lead ECG showing the following: having a corrected QTc interval > 450 msec or <320 msec (Fridericia's correction);
* sustained sitting systolic blood pressure > 140 or < 90 mm Hg or sitting diastolic blood pressure > 90 or < 50 mm Hg at Screening or Day -1 (sentinel pair) or Day 1 (remaining 6 subjects in the cohort), the average of the 2 assessments of BP taken at each visit will be used to exclude a subject;
* resting pulse rate at screening of > 100 or < 45;
* donated or lost > 500 mL of blood < 56 days prior to enrollment into this study;
* plasma donation within 7 days prior to enrollment into this study;
* active infection or febrile illness < 14 days prior to the first dose of study medication;
* use of prescription or over-the-counter medications or herbal supplements ≤ 14 days prior to dosing and until completion of follow-up visit on Day 7;
* have participated in other clinical studies of a new chemical entity within 30 days prior to admission to the CRU.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety, including adverse events, physical examinations, ECGs, clinical laboratory tests | Screening (28 days prior to dosing) through Day 7
  Safety, as determined by the number of participants with adverse events related to treatment, the number of participants with clinically significant changes in blood pressure, heart rate and respiration, the number of participants with abnormal laboratory values, the number of participants with abnormal ECGs.

SECONDARY OUTCOMES:
To possibly determine the maximally tolerated dose (MTD) of orally administered NPT200-11 in healthy subjects. | Screening (28 days prior to dosing) through Day 7 of MTD
  The number of participants with unacceptable toxicities at each dose level will determine the maximally tolerated dose.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, M.D. CPI, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States